CLINICAL TRIAL: NCT07072793
Title: Work Productivity Losses in the United States Among High-risk Patients With COVID-19 During Acute and Longer-term Follow-up in an Omicron Predominant Period (PULSE-US)
Brief Title: A US Study to Look at Loss of Work and Healthcare Costs for People Affected With Mild-to-moderate COVID 19 Who Have High Chances of the Disease Becoming Severe
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C4671066
Record Dates: First submitted 2024-11-15; First posted 2025-07-18 (Actual); Results first posted 2026-01-12 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: COVID-19 (Coronavirus Disease 2019)
Keywords: SARS Coronavirus; SARS Virus; SARS-CoV; SARS-CoV-1; Paxlovid; omicron
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome | interventions — nirmatrelvir and ritonavir drug combination

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Treated cohort: nirmatrelvir-ritonavir: Participants with confirmed diagnosis of Covid-19 and with mild to moderate symptoms at high-risk for progressing to severe disease.
  Interventions: Drug: nirmatrelvir-ritonavir
- Untreated cohort: not receiving any antiviral treatment: Participants with confirmed diagnosis of Covid-19 and with mild to moderate symptoms at high-risk for progressing to severe disease.

INTERVENTIONS:
Drug: nirmatrelvir-ritonavir — Participants with confirmed diagnosis of Covid-19 and with mild to moderate symptoms at high-risk for progressing to severe disease
  Other Names: Paxlovid
  Groups: Treated cohort: nirmatrelvir-ritonavir

SUMMARY:
The purpose of this study is to understand how COVID-19 affects people's ability to work and to calculate the costs associated with loss of work.

The study compares two groups of participants who are confirmed to have mild-to moderated COVID-19 and who have high chances of the disease becoming severe.

The two groups are:

People who took the antiviral medication nirmatrelvir-ritonavir (also called Paxlovid) People who were eligible to receive antiviral medication but did not receive any.

The participants will be selected from various health databases in the US between June 2021 and December 2022.

The main goals are:

To look at the characteristics of both groups of participants with COVID-19. To measure how much work these participants missed, including days off and sick leave, and the costs associated with this work loss.

To compare work loss and costs between the two groups of participants, considering differences in their clinical and demographic characteristics.

The study will evaluate at least 30 days of data from participants after they are confirmed to have COVID-19

ELIGIBILITY:
Inclusion Criteria:

* >1 non-diagnostic2 outpatient medical claim in the MarketScan Commercial or Medicare Database with the International Classification of Diseases, 10th Revision (ICD-10) diagnosis code for COVID-19 (U071) between December 16, 2021 (5 days prior to the date of emergency use authorization of NMV/r) and December 1, 2022 (30 days prior to the end of available HPM data); the date of the earliest qualifying claim is the index date.
* Primary beneficiary on their insurance policy (i.e., eligible for inclusion in the MarketScan HPM Database)
* >6 months of continuous enrollment with medical and pharmacy benefits in the MarketScan Commercial or Medicare Database before the index date (baseline period)
* >30 days of continuous enrollment with medical and pharmacy benefits in the MarketScan Commercial or Medicare Database after and including the index date (minimum follow-up period)
* Treated cohort ONLY: ≥1 claim for Paxlovid within 5 days of index (index date and next 4 days)

Exclusion Criteria:

* Evidence of death on the index date or the following day
* Any inpatient admission on the index date or the following day
* ≥1 inpatient claim with a COVID-19 diagnosis in any position on the claim during the 30 days before the index date
* >1 non-diagnostic claim with a diagnosis code for stage 4 or stage 5 chronic kidney disease, end stage renal disease, or a procedure code for dialysis, during the baseline period or on the index date

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: retrospective cohort study of adult, high-risk patients diagnosed with COVID-19 using data from the Merative™ MarketScan® Commercial, Medicare, and Health and Productivity Management (HPM) Databases. The index date for both cohorts will be the date of the first COVID-19 diagnosis and patients will be followed over a 6-month pre-period and variable post-period. The post-period will be a minimum of 30 days to allow patients the opportunity to experience the primary study outcomes of work loss days (absence, STD, and LTD) along with associated indirect costs.
Sampling Method: Non-Probability Sample
Enrollment: 131005 (Actual)
Dates: Start 2024-10-31 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2024-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer New York, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4671066

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data of eligible participants in the US diagnosed with coronavirus disease 2019 (COVID-19) who received nirmatrelvir-ritonavir (NMV/r) [Paxlovid] or did not receive any antiviral therapy for COVID-19 was included in this retrospective observational study. In this study, outcome measures were evaluated for actual enrolled numbers (unmatched population) and matched numbers (pseudo population) derived by matching pre-defined characteristics among actual enrolled numbers.
Pre-assignment Details: Participants with COVID-19 diagnosis from 16-Dec-2021 to 1-Dec-2022 (approx. 11.5 months of index date identification period) were identified to be included in study. Data was retrieved from 19-Jun-2021 to 31-Dec-2022 (approx. 1.5 years) using the Merative™ MarketScan® database (Commercial and Medicare participants; Health and Productivity Management [HPM] database). Data was evaluated per study objectives, from 31-Oct-2024 (study start) to 15-Nov-2024 (study completion) [approx. 0.5 months].
Groups:
- Unmatched Treated Cohort: Participants who were diagnosed with COVID-19 and had received NMV/r for COVID-19 were included in this cohort. Their data was studied retrospectively. No intervention was administered in this study. This arm contains participants who were not matched for any pre-defined characteristics and are the actual enrolled numbers.
- Unmatched Untreated Cohort: Participants who were diagnosed with COVID-19 and did not receive any antiviral therapy for COVID-19 were included in this cohort. Their data was studied retrospectively. This arm contains participants who were not matched for pre-defined characteristics and are the actual enrolled numbers.
Period: Overall Study
Arm/Group | Unmatched Treated Cohort | Unmatched Untreated Cohort
Started (Actual enrolled number) | 23155 (Actual enrolled number) | 107850 (Actual enrolled number)
Completed | 23155 | 107850
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all eligible participants whose data was retrieved and observed in this study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Unmatched Treated Cohort | Unmatched Untreated Cohort | Total
Number analyzed (Participants) | 23155 | 107850 | 131005
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23062 | 107708 | 130770
  >=65 years | 93 | 142 | 235
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11156 | 52578 | 63734
  Male | 11999 | 55272 | 67271
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants According to Age Group: Unmatched Participants
Description: Age group was categorized into following categories: 18-29 years, 30-39 years, 40-49 years, 50-64 years and 65-74 years. Index date was the date of first COVID-19 diagnosis. In this outcome measure, data was reported for unmatched participants, they were further sub-grouped on the basis of outcome of COVID-19: eligible for absence from work, eligible for short term disability and eligible for long term disability. These sub-groups were not mutually exclusive; some participants might be represented in more than one category.
Time Frame: At index date (any date during index date identification period of approximately 11.5 months); retrospective data collected was evaluated in 0.5 months of this study
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study. This outcome measure was planned to be reported for unmatched participants (treated and untreated).
Measure: Count of Participants; unit: Participants
Groups:
- Unmatched Treated: Absence Eligibility: Participants who received NMV/r for COVID-19 and were eligible for absence from work, were included in this cohort. This arm contains participants who were not matched for any pre-defined characteristics and are the actual numbers.
- Unmatched Untreated: Absence Eligibility: Participants who did not receive any antiviral therapy for COVID-19 and were eligible for absence from work, were included in this cohort. This arm contains participants who were not matched for any pre-defined characteristics and are the actual numbers.
- Unmatched Treated: Short-term Disability: Participants who received NMV/r for COVID-19 and were eligible for short term disability, were included in this cohort. This arm contains participants who were not matched for any pre-defined characteristics and are the actual numbers.
- Unmatched Untreated: Short-term Disability: Participants who did not receive any antiviral therapy for COVID-19 and were eligible for short term disability, were included in this cohort. This arm contains participants who were not matched for any pre-defined characteristics and are the actual numbers.
- Unmatched Treated: Long-term Disability: Participants who received NMV/r for COVID-19 and were eligible for long term disability, were included in this cohort. This arm contains participants who were not matched for any pre-defined characteristics and are the actual numbers.
- Unmatched Untreated: Long-term Disability: Participants who did not receive any antiviral therapy for COVID-19 and were eligible for long term disability, were included in this cohort. This arm contains participants who were not matched for any pre-defined characteristics and are the actual numbers.
Arm/Group | Unmatched Treated: Absence Eligibility | Unmatched Untreated: Absence Eligibility | Unmatched Treated: Short-term Disability | Unmatched Untreated: Short-term Disability | Unmatched Treated: Long-term Disability | Unmatched Untreated: Long-term Disability
Number analyzed (Participants) | 1931 | 9092 | 20076 | 90459 | 20336 | 94818
Participants
  18-29 years | 57 | 686 | 545 | 6123 | 556 | 6493
  30-39 years | 201 | 1442 | 2076 | 15168 | 2087 | 16006
  40-49 years | 349 | 1926 | 3862 | 19715 | 3850 | 20271
  50-64 years | 1271 | 4850 | 12971 | 47814 | 13180 | 50312
  65-74 years | 53 | 188 | 622 | 1639 | 663 | 1736

2. Primary Outcome: Number of Participants According to Age Group: Matched Participants
Description: Age group was categorized into following categories: 18-29 years, 30-39 years, 40-49 years, 50-64 years and 65-74 years. Index date was the date of first COVID-19 diagnosis. In this outcome measure, data was reported for matched participants, they were further sub-grouped on the basis of outcome of COVID-19: eligible for absence from work, eligible for short term disability and eligible for long term disability. These sub-groups were not mutually exclusive; some participants might be represented in more than one category.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study. This outcome measure was planned to be reported for matched participants (treated and untreated). Here, "Overall Number of Participants Analyzed" signifies the numbers which were matched/ adjusted based on pre-defined characteristics among actual enrolled population and was a pseudo population, hence these numbers are different from unmatched population (actual enrolled population).
Measure: Count of Participants; unit: Participants
Groups:
- Matched Treated: Absence Eligibility: Participants who received NMV/r for COVID-19 and were eligible for absence from work, were included in this cohort. This arm contains participants who were matched for pre-defined characteristics and are the matched/ adjusted numbers.
- Matched Untreated: Absence Eligibility: Participants who did not receive any antiviral therapy for COVID-19 and were eligible for absence from work, were included in this cohort. This arm contains participants who were matched for pre-defined characteristics and are the matched/ adjusted numbers.
- Matched Treated: Short-term Disability: Participants who received NMV/r for COVID-19 and were eligible for short term disability, were included in this cohort. This arm contains participants who were matched for pre-defined characteristics and are the matched/ adjusted numbers.
- Matched Untreated: Short-term Disability: Participants who did not receive any antiviral therapy for COVID-19 and were eligible for short term disability, were included in this cohort. This arm contains participants who were matched for pre-defined characteristics and are the matched/ adjusted numbers.
- Matched Treated: Long-term Disability: Participants who received NMV/r for COVID-19 and were eligible for long term disability, were included in this cohort. This arm contains participants who were matched for pre-defined characteristics and are the matched/ adjusted numbers.
- Matched Untreated: Long-term Disability: Participants who did not receive any antiviral therapy for COVID-19 and were eligible for long term disability, were included in this cohort. This arm contains participants who were matched for pre-defined characteristics and are the matched/ adjusted numbers.
Arm/Group | Matched Treated: Absence Eligibility | Matched Untreated: Absence Eligibility | Matched Treated: Short-term Disability | Matched Untreated: Short-term Disability | Matched Treated: Long-term Disability | Matched Untreated: Long-term Disability
Number analyzed (Participants) | 1909 | 1909 | 20065 | 20065 | 20318 | 20318
Participants
  18-29 years | 56 | 63 | 543 | 541 | 554 | 553
  30-39 years | 199 | 197 | 2076 | 2081 | 2087 | 2094
  40-49 years | 345 | 349 | 3862 | 3727 | 3850 | 3738
  50-64 years | 1258 | 1248 | 12963 | 13271 | 13172 | 13469
  65-74 years | 51 | 52 | 621 | 445 | 655 | 464

3. Primary Outcome: Number of Participants According to Sex: Unmatched Participants
Description: Sex was categorized as: female and male. Index date was the date of first COVID-19 diagnosis. In this outcome measure, data was reported for unmatched participants, they were further sub-grouped on the basis of outcome of COVID-19: eligible for absence from work, eligible for short term disability and eligible for long term disability. These sub-groups were not mutually exclusive; some participants might be represented in more than one category.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Unmatched Treated: Absence Eligibility | Unmatched Untreated: Absence Eligibility | Unmatched Treated: Short-term Disability | Unmatched Untreated: Short-term Disability | Unmatched Treated: Long-term Disability | Unmatched Untreated: Long-term Disability
Number analyzed (Participants) | 1931 | 9092 | 20076 | 90459 | 20336 | 94818
Participants
  Female | 923 | 3991 | 9466 | 42650 | 9916 | 46815
  Male | 1008 | 5101 | 10610 | 47809 | 10420 | 48003

4. Primary Outcome: Number of Participants According to Sex: Matched Participants
Description: Sex was categorized as: female and male. Index date was the date of first COVID-19 diagnosis. In this outcome measure, data was reported for matched participants, they were further sub-grouped on the basis of outcome of COVID-19: eligible for absence from work, eligible for short term disability and eligible for long term disability. These sub-groups were not mutually exclusive; some participants might be represented in more than one category.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Matched Treated: Absence Eligibility | Matched Untreated: Absence Eligibility | Matched Treated: Short-term Disability | Matched Untreated: Short-term Disability | Matched Treated: Long-term Disability | Matched Untreated: Long-term Disability
Number analyzed (Participants) | 1909 | 1909 | 20065 | 20065 | 20318 | 20318
Participants
  Female | 914 | 914 | 9462 | 9462 | 9916 | 9916
  Male | 995 | 995 | 10603 | 10603 | 10402 | 10402

5. Primary Outcome: Number of Participants According to Region of Residence: Unmatched Participants
Description: Region of residence was categorized into following categories: Northeast, North Central, South, West, and other/ missing. Index date was the date of first COVID-19 diagnosis. In this outcome measure, data was reported for unmatched participants, they were further sub-grouped on the basis of outcome of COVID-19: eligible for absence from work, eligible for short term disability and eligible for long term disability. These sub-groups were not mutually exclusive; some participants might be represented in more than one category.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Unmatched Treated: Absence Eligibility | Unmatched Untreated: Absence Eligibility | Unmatched Treated: Short-term Disability | Unmatched Untreated: Short-term Disability | Unmatched Treated: Long-term Disability | Unmatched Untreated: Long-term Disability
Number analyzed (Participants) | 1931 | 9092 | 20076 | 90459 | 20336 | 94818
Participants
  Northeast | 120 | 657 | 3335 | 13377 | 3386 | 13012
  North Central | 703 | 2597 | 4184 | 21364 | 4598 | 24047
  South | 955 | 5127 | 7903 | 41391 | 7567 | 43011
  West | 153 | 708 | 4634 | 14130 | 4765 | 14552
  Other/missing | 0 | 3 | 20 | 197 | 20 | 196

6. Primary Outcome: Number of Participants According to Region of Residence: Matched Participants
Description: Region of residence was categorized into following categories: Northeast, North Central, South, West and other/ missing. Index date was the date of first COVID-19 diagnosis. In this outcome measure, data was reported for matched participants, they were further sub-grouped on the basis of outcome of COVID-19: eligible for absence from work, eligible for short term disability and eligible for long term disability. These sub-groups were not mutually exclusive; some participants might be represented in more than one category.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Matched Treated: Absence Eligibility | Matched Untreated: Absence Eligibility | Matched Treated: Short-term Disability | Matched Untreated: Short-term Disability | Matched Treated: Long-term Disability | Matched Untreated: Long-term Disability
Number analyzed (Participants) | 1909 | 1909 | 20065 | 20065 | 20318 | 20318
Participants
  Northeast | 119 | 140 | 3332 | 3258 | 3381 | 3044
  North Central | 694 | 602 | 4180 | 4755 | 4592 | 5045
  South | 944 | 994 | 7902 | 8376 | 7563 | 8551
  West | 152 | 173 | 4631 | 3620 | 4762 | 3614
  Other/missing | 0 | 0 | 20 | 56 | 20 | 64

7. Primary Outcome: Number of Participants According to Payer Type: Unmatched Participants
Description: Payer type was categorized as: commercial and medicare. Index date was the date of first COVID-19 diagnosis. In this outcome measure, data was reported for unmatched participants, they were further sub-grouped on the basis of outcome of COVID-19: eligible for absence from work, eligible for short term disability and eligible for long term disability. These sub-groups were not mutually exclusive; some participants might be represented in more than one category.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were included and observed in this study. This outcome measure was planned to be reported for unmatched participants (treated and untreated).
Measure: Count of Participants; unit: Participants
Arm/Group | Unmatched Treated: Absence Eligibility | Unmatched Untreated: Absence Eligibility | Unmatched Treated: Short-term Disability | Unmatched Untreated: Short-term Disability | Unmatched Treated: Long-term Disability | Unmatched Untreated: Long-term Disability
Number analyzed (Participants) | 1931 | 9092 | 20076 | 90459 | 20336 | 94818
Participants
  Commercial | 1923 | 9082 | 20005 | 90353 | 20261 | 94703
  Medicare | 8 | 10 | 71 | 106 | 75 | 115

8. Primary Outcome: Number of Participants According to Payer Type: Matched Participants
Description: Payer type was categorized as: commercial and medicare. Index date was the date of first COVID-19 diagnosis. In this outcome measure, data was reported for matched participants, they were further sub-grouped on the basis of outcome of COVID-19: eligible for absence from work, eligible for short term disability and eligible for long term disability. These sub-groups were not mutually exclusive; some participants might be represented in more than one category.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Matched Treated: Absence Eligibility | Matched Untreated: Absence Eligibility | Matched Treated: Short-term Disability | Matched Untreated: Short-term Disability | Matched Treated: Long-term Disability | Matched Untreated: Long-term Disability
Number analyzed (Participants) | 1909 | 1909 | 20065 | 20065 | 20318 | 20318
Participants
  Commercial | 1902 | 1907 | 19994 | 20013 | 20245 | 20270
  Medicare | 7 | 2 | 71 | 52 | 73 | 48

9. Primary Outcome: Number of Participants According to Insurance Plan Type: Unmatched Participants
Description: Insurance plan type was categorized into following categories: comprehensive/indemnity, exclusive/preferred provider organization (EPO/PPO), point of service capitation (POS) with or without capitation, health maintenance organization (HMO), consumer driven/ high-deductible health plan (CDHP/HDHP) and missing/unknown. Index date was the date of first COVID-19 diagnosis. In this outcome measure, data was reported for unmatched participants, they were further sub-grouped on the basis of outcome of COVID-19: eligible for absence from work, eligible for short term disability and eligible for long term disability. These sub-groups were not mutually exclusive; some participants might be represented in more than one category.
Time Frame: as for outcome 1
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Unmatched Treated: Absence Eligibility | Unmatched Untreated: Absence Eligibility | Unmatched Treated: Short-term Disability | Unmatched Untreated: Short-term Disability | Unmatched Treated: Long-term Disability | Unmatched Untreated: Long-term Disability
Number analyzed (Participants) | 1931 | 9092 | 20076 | 90459 | 20336 | 94818
Participants
  Comprehensive/indemnity | 12 | 73 | 722 | 2637 | 381 | 3277
  EPO/PPO | 444 | 2332 | 7433 | 35597 | 8692 | 44960
  POS with or without capitation | 2 | 32 | 236 | 1093 | 362 | 1642
  HMO | 446 | 1637 | 2452 | 9662 | 2865 | 10903
  CDHP/HDHP | 1021 | 4996 | 8923 | 40222 | 7720 | 32766
  Missing/unknown | 6 | 22 | 310 | 1248 | 316 | 1270

10. Primary Outcome: Number of Participants According to Insurance Plan Type: Matched Participants
Description: Insurance plan type was categorized into following categories: comprehensive/indemnity, EPO/PPO, POS with or without capitation, HMO, CDHP/HDHP and missing/unknown. Index date was the date of first COVID-19 diagnosis. In this outcome measure, data was reported for matched participants, they were further sub-grouped on the basis of outcome of COVID-19: eligible for absence from work, eligible for short term disability and eligible for long term disability. These sub-groups were not mutually exclusive; some participants might be represented in more than one category.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Matched Treated: Absence Eligibility | Matched Untreated: Absence Eligibility | Matched Treated: Short-term Disability | Matched Untreated: Short-term Disability | Matched Treated: Long-term Disability | Matched Untreated: Long-term Disability
Number analyzed (Participants) | 1909 | 1909 | 20065 | 20065 | 20318 | 20318
Participants
  Comprehensive/indemnity | 12 | 19 | 721 | 601 | 380 | 548
  EPO/PPO | 439 | 485 | 7430 | 8228 | 8683 | 9849
  POS with or without capitation | 2 | 1 | 236 | 272 | 362 | 356
  HMO | 442 | 377 | 2450 | 2242 | 2863 | 2437
  CDHP/HDHP | 1008 | 1022 | 8918 | 8439 | 7714 | 6859
  Missing/unknown | 6 | 5 | 310 | 283 | 316 | 269

11. Primary Outcome: Number of Participants According to Industry Type: Unmatched Participants
Description: Industry type was categorized into following categories: finance/insurance/real estate, manufacturing (durable/non-durable goods), retail trade, services, transportation/communications/utilities and other. Index date was the date of first COVID-19 diagnosis. In this outcome measure, data was reported for unmatched participants, they were further sub-grouped on the basis of outcome of COVID-19: eligible for absence from work, eligible for short term disability and eligible for long term disability. These sub-groups were not mutually exclusive; some participants might be represented in more than one category.
Time Frame: as for outcome 1
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Unmatched Treated: Absence Eligibility | Unmatched Untreated: Absence Eligibility | Unmatched Treated: Short-term Disability | Unmatched Untreated: Short-term Disability | Unmatched Treated: Long-term Disability | Unmatched Untreated: Long-term Disability
Number analyzed (Participants) | 1931 | 9092 | 20076 | 90459 | 20336 | 94818
Participants
  Finance/insurance/real estate | 0 | 0 | 3352 | 13278 | 3414 | 13003
  Manufacturing (durable goods) | 440 | 1949 | 5463 | 27791 | 4713 | 27153
  Manufacturing (non-durable goods) | 0 | 0 | 2157 | 10527 | 2171 | 10619
  Retail trade | 0 | 0 | 764 | 3754 | 783 | 3853
  Services | 506 | 1562 | 3340 | 11964 | 4808 | 16470
  Transportation/communications/utilities | 985 | 5581 | 3114 | 17433 | 2402 | 13235
  Other | 0 | 0 | 1886 | 5712 | 2045 | 10485

12. Primary Outcome: Number of Participants According to Industry Type: Matched Participants
Description: Industry type was categorized into following categories: finance/insurance/real estate, manufacturing (durable/non-durable goods), retail trade, services, transportation/communications/utilities and other. Index date was the date of first COVID-19 diagnosis. In this outcome measure, data was reported for matched participants, they were further sub-grouped on the basis of outcome of COVID-19: eligible for absence from work, eligible for short term disability and eligible for long term disability. These sub-groups were not mutually exclusive; some participants might be represented in more than one category.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Matched Treated: Absence Eligibility | Matched Untreated: Absence Eligibility | Matched Treated: Short-term Disability | Matched Untreated: Short-term Disability | Matched Treated: Long-term Disability | Matched Untreated: Long-term Disability
Number analyzed (Participants) | 1909 | 1909 | 20065 | 20065 | 20318 | 20318
Participants
  Finance/insurance/real estate | 0 | 0 | 3351 | 2729 | 3411 | 2673
  Manufacturing (durable goods) | 435 | 406 | 5459 | 6257 | 4707 | 5643
  Manufacturing (non-durable goods) | 0 | 0 | 2155 | 2262 | 2169 | 2226
  Retail trade | 0 | 0 | 764 | 783 | 783 | 769
  Services | 501 | 386 | 3339 | 2931 | 4806 | 3815
  Transportation/communications/utilities | 973 | 1117 | 3112 | 3414 | 2400 | 2481
  Other | 0 | 0 | 1885 | 1689 | 2042 | 2711

13. Primary Outcome: Number of Participants According to Quarter (Q) of Index Year: Unmatched Participants
Description: Quarter of index year was categorized into following categories: Q4 2021, Q1 2022, Q2 2022, Q3 2022 and Q4 2022. Index date was the date of first COVID-19 diagnosis. In this outcome measure, data was reported for unmatched participants, they were further sub-grouped on the basis of outcome of COVID-19: eligible for absence from work, eligible for short term disability and eligible for long term disability. These sub-groups were not mutually exclusive; some participants might be represented in more than one category.
Time Frame: as for outcome 1
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Unmatched Treated: Absence Eligibility | Unmatched Untreated: Absence Eligibility | Unmatched Treated: Short-term Disability | Unmatched Untreated: Short-term Disability | Unmatched Treated: Long-term Disability | Unmatched Untreated: Long-term Disability
Number analyzed (Participants) | 1931 | 9092 | 20076 | 90459 | 20336 | 94818
Participants
  Q4 2021 | 1 | 1255 | 3 | 10991 | 3 | 11766
  Q1 2022 | 23 | 3587 | 132 | 33169 | 127 | 34383
  Q2 2022 | 523 | 1705 | 5720 | 17345 | 5842 | 18233
  Q3 2022 | 1037 | 1909 | 10424 | 21706 | 10502 | 22854
  Q4 2022 | 347 | 636 | 3797 | 7248 | 3862 | 7582

14. Primary Outcome: Number of Participants According to Quarter of Index Year: Matched Participants
Description: Quarter of index year was categorized into following categories: Q4 2021, Q1 2022, Q2 2022, Q3 2022 and Q4 2022. Index date was the date of first COVID-19 diagnosis. In this outcome measure, data was reported for matched participants, they were further sub-grouped on the basis of outcome of COVID-19: eligible for absence from work, eligible for short term disability and eligible for long term disability. These sub-groups were not mutually exclusive; some participants might be represented in more than one category.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Matched Treated: Absence Eligibility | Matched Untreated: Absence Eligibility | Matched Treated: Short-term Disability | Matched Untreated: Short-term Disability | Matched Treated: Long-term Disability | Matched Untreated: Long-term Disability
Number analyzed (Participants) | 1909 | 1909 | 20065 | 20065 | 20318 | 20318
Participants
  Q4 2021 | 1 | 1 | 3 | 3 | 3 | 3
  Q1 2022 | 23 | 23 | 132 | 132 | 127 | 127
  Q2 2022 | 520 | 520 | 5720 | 5720 | 5842 | 5842
  Q3 2022 | 1028 | 1028 | 10424 | 10424 | 10502 | 10502
  Q4 2022 | 337 | 337 | 3786 | 3786 | 3844 | 3844

15. Primary Outcome: Mean Duration of Follow-up: Unmatched Participants
Description: Duration of follow-up was defined as number of months from (and including) the index date to the end of participants variable-length follow-up period. Index date was the date of first COVID-19 diagnosis. In this outcome measure, data was reported for unmatched participants, they were further sub-grouped on the basis of outcome of COVID-19: eligible for absence from work, eligible for short term disability and eligible for long term disability. These sub-groups were not mutually exclusive; some participants might be represented in more than one category.
Time Frame: From index date to the end of follow-up (maximum follow-up was up to an average of 8.3 months during data observation of approximately 1.5 years); retrospective data collected was evaluated in 0.5 months of this study
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Unmatched Treated: Absence Eligibility | Unmatched Untreated: Absence Eligibility | Unmatched Treated: Short-term Disability | Unmatched Untreated: Short-term Disability | Unmatched Treated: Long-term Disability | Unmatched Untreated: Long-term Disability
Number analyzed (Participants) | 1931 | 9092 | 20076 | 90459 | 20336 | 94818
Months | 4.9 (2.0) | 8.3 (3.6) | 4.9 (2.0) | 8.0 (3.6) | 4.9 (2.0) | 8.0 (3.6)

16. Primary Outcome: Mean Duration of Follow-up: Matched Participants
Description: Duration of follow-up was defined as number of months from (and including) the index date to the end of participants variable-length follow-up period. Index date was the date of first COVID-19 diagnosis. In this outcome measure, data was reported for matched participants, they were further sub-grouped on the basis of outcome of COVID-19: eligible for absence from work, eligible for short term disability and eligible for long term disability. These sub-groups were not mutually exclusive; some participants might be represented in more than one category.
Time Frame: as for outcome 15
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Matched Treated: Absence Eligibility | Matched Untreated: Absence Eligibility | Matched Treated: Short-term Disability | Matched Untreated: Short-term Disability | Matched Treated: Long-term Disability | Matched Untreated: Long-term Disability
Number analyzed (Participants) | 1909 | 1909 | 20065 | 20065 | 20318 | 20318
Months | 4.9 (2.0) | 5.0 (2.1) | 4.9 (2.0) | 5.0 (2.1) | 4.9 (2.0) | 5.0 (2.1)

17. Primary Outcome: Mean Elixhauser Comorbidity Index (ECI): Unmatched Participants
Description: ECI was a measure of comorbidity based on ICD-10 codes. ECI score range was from 0-30. A higher score indicated more comorbidity. Index date was the date of first COVID-19 diagnosis. In this outcome measure, data was reported for unmatched participants, they were further sub-grouped on the basis of outcome of COVID-19: eligible for absence from work, eligible for short term disability and eligible for long term disability. These sub-groups were not mutually exclusive; some participants might be represented in more than one category.
Time Frame: Pre-period (6 months period before index date; during data observation of approximately 1.5 years); retrospective data collected was evaluated in 0.5 months of this study
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Unmatched Treated: Absence Eligibility | Unmatched Untreated: Absence Eligibility | Unmatched Treated: Short-term Disability | Unmatched Untreated: Short-term Disability | Unmatched Treated: Long-term Disability | Unmatched Untreated: Long-term Disability
Number analyzed (Participants) | 1931 | 9092 | 20076 | 90459 | 20336 | 94818
Units on a scale | 1.3 (1.2) | 1.2 (1.2) | 1.3 (1.2) | 1.2 (1.2) | 1.3 (1.2) | 1.2 (1.2)

18. Primary Outcome: Mean ECI: Matched Participants
Description: ECI was a measure of comorbidity based on ICD-10 codes. ECI score range was from 0-30. A higher score indicated more comorbidity. Index date was the date of first COVID-19 diagnosis. In this outcome measure, data was reported for matched participants, they were further sub-grouped on the basis of outcome of COVID-19: eligible for absence from work, eligible for short term disability and eligible for long term disability. These sub-groups were not mutually exclusive; some participants might be represented in more than one category.
Time Frame: as for outcome 17
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Matched Treated: Absence Eligibility | Matched Untreated: Absence Eligibility | Matched Treated: Short-term Disability | Matched Untreated: Short-term Disability | Matched Treated: Long-term Disability | Matched Untreated: Long-term Disability
Number analyzed (Participants) | 1909 | 1909 | 20065 | 20065 | 20318 | 20318
Units on a scale | 1.3 (1.2) | 1.2 (1.2) | 1.3 (1.2) | 1.2 (1.2) | 1.3 (1.2) | 1.2 (1.2)

19. Primary Outcome: Mean Charlson Comorbidity Index (CCI): Unmatched Participants
Description: CCI based on various comorbid conditions such as cerebrovascular disease, chronic pulmonary disease, congestive heart failure, dementia, mild/moderate diabetes, diabetes with chronic complications, hemiplegia/paraplegia, human immunodeficiency virus(HIV), mild liver disease, moderate/severe liver disease, malignancy, metastatic solid tumor, myocardial infarction, peptic ulcer disease, peripheral vascular disease, renal disease, rheumatologic disease was reported. CCI score range was from 0 to 33, where "0"= low comorbid condition and "33"= high comorbid condition, higher scores indicated more comorbidity. Index date was the date of first COVID-19 diagnosis. Data was reported for unmatched participants, they were further sub-grouped on the basis of outcome of COVID-19: eligible for absence from work, eligible for short term disability and eligible for long term disability. These sub-groups were not mutually exclusive; some participants might be represented in more than one category.
Time Frame: as for outcome 17
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Unmatched Treated: Absence Eligibility | Unmatched Untreated: Absence Eligibility | Unmatched Treated: Short-term Disability | Unmatched Untreated: Short-term Disability | Unmatched Treated: Long-term Disability | Unmatched Untreated: Long-term Disability
Number analyzed (Participants) | 1931 | 9092 | 20076 | 90459 | 20336 | 94818
Units on a scale | 0.6 (1.1) | 0.6 (1.2) | 0.7 (1.2) | 0.6 (1.1) | 0.7 (1.2) | 0.6 (1.1)

20. Primary Outcome: Mean CCI: Matched Participants
Description: CCI based on various comorbid conditions such as cerebrovascular disease, chronic pulmonary disease, congestive heart failure, dementia, mild/moderate diabetes, diabetes with chronic complications, hemiplegia/paraplegia, HIV, mild liver disease, moderate/severe liver disease, malignancy, metastatic solid tumor, myocardial infarction, peptic ulcer disease, peripheral vascular disease, renal disease, rheumatologic disease was reported. CCI score range was from 0 to 33, where "0"= low comorbid condition and "33"= high comorbid condition, higher scores indicated more comorbidity. Index date was the date of first COVID-19 diagnosis. In this outcome measure, data was reported for matched participants, they were further sub-grouped on the basis of outcome of COVID-19: eligible for absence from work, eligible for short term disability and eligible for long term disability. These sub-groups were not mutually exclusive; some participants might be represented in more than one category.
Time Frame: as for outcome 17
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Matched Treated: Absence Eligibility | Matched Untreated: Absence Eligibility | Matched Treated: Short-term Disability | Matched Untreated: Short-term Disability | Matched Treated: Long-term Disability | Matched Untreated: Long-term Disability
Number analyzed (Participants) | 1909 | 1909 | 20065 | 20065 | 20318 | 20318
Units on a scale | 0.6 (1.1) | 0.6 (1.1) | 0.7 (1.2) | 0.6 (1.2) | 0.7 (1.2) | 0.6 (1.2)

21. Primary Outcome: Number of Participants According to Comorbidities: Unmatched Participants
Description: Comorbidities were categorized into following categories: cancer (current or history of), cardio/cerebrovascular disease, chronic kidney disease, chronic liver disease, diabetes mellitus, immunocompromised status, lung disease or tuberculosis, neurodevelopmental disorder/complex condition, overweight/obesity or smoking and pregnancy. Index date was the date of first COVID-19 diagnosis. In this outcome measure, data was reported for unmatched participants, they were further sub-grouped on the basis of outcome of COVID-19: eligible for absence from work, eligible for short term disability and eligible for long term disability. These sub-groups were not mutually exclusive; some participants might be represented in more than one category. Participant can have more than 1 comorbidity.
Time Frame: as for outcome 17
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Unmatched Treated: Absence Eligibility | Unmatched Untreated: Absence Eligibility | Unmatched Treated: Short-term Disability | Unmatched Untreated: Short-term Disability | Unmatched Treated: Long-term Disability | Unmatched Untreated: Long-term Disability
Number analyzed (Participants) | 1931 | 9092 | 20076 | 90459 | 20336 | 94818
Participants
  Cancer (current or history of) | 156 | 607 | 1796 | 6307 | 1817 | 6596
  Cardio/cerebrovascular disease | 690 | 2969 | 7032 | 28860 | 6959 | 30181
  Chronic kidney disease | 19 | 106 | 165 | 789 | 158 | 801
  Chronic liver disease | 37 | 142 | 391 | 1507 | 362 | 1495
  Diabetes mellitus | 280 | 1042 | 3143 | 10280 | 3115 | 10565
  Immunocompromised status | 365 | 1985 | 3448 | 16695 | 3508 | 17543
  Lung disease or tuberculosis | 78 | 383 | 828 | 3716 | 849 | 3920
  Neurodevelopmental disorder/complex condition | 372 | 1767 | 3683 | 18640 | 3805 | 19761
  Overweight/obesity or smoking | 696 | 3329 | 6680 | 31046 | 6699 | 32689
  Pregnancy | 18 | 291 | 193 | 3108 | 209 | 3414

22. Primary Outcome: Number of Participants According to Comorbidities: Matched Participants
Description: Comorbidities were categorized into following categories: cancer (current or history of), cardio/cerebrovascular disease, chronic kidney disease, chronic liver disease, diabetes mellitus, immunocompromised status, lung disease or tuberculosis, neurodevelopmental disorder/complex condition, overweight/obesity or smoking and pregnancy. Index date was the date of first COVID-19 diagnosis. In this outcome measure, data was reported for matched participants, they were further sub-grouped on the basis of outcome of COVID-19: eligible for absence from work, eligible for short term disability and eligible for long term disability. These sub-groups were not mutually exclusive; some participants might be represented in more than one category. Participant can have more than 1 comorbidity.
Time Frame: as for outcome 17
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Matched Treated: Absence Eligibility | Matched Untreated: Absence Eligibility | Matched Treated: Short-term Disability | Matched Untreated: Short-term Disability | Matched Treated: Long-term Disability | Matched Untreated: Long-term Disability
Number analyzed (Participants) | 1909 | 1909 | 20065 | 20065 | 20318 | 20318
Participants
  Cancer (current or history of) | 150 | 132 | 1792 | 1677 | 1811 | 1665
  Cardio/cerebrovascular disease | 677 | 634 | 7026 | 6603 | 6948 | 6670
  Chronic kidney disease | 17 | 22 | 165 | 221 | 157 | 212
  Chronic liver disease | 37 | 23 | 391 | 355 | 372 | 330
  Diabetes mellitus | 269 | 218 | 3139 | 2555 | 3103 | 2478
  Immunocompromised status | 356 | 370 | 3445 | 3281 | 3504 | 3376
  Lung disease or tuberculosis | 77 | 67 | 826 | 779 | 847 | 810
  Neurodevelopmental disorder/complex condition | 376 | 357 | 3780 | 3732 | 3802 | 3733
  Overweight/obesity or smoking | 683 | 658 | 6675 | 6164 | 6692 | 6257
  Pregnancy | 18 | 38 | 193 | 409 | 209 | 437

23. Primary Outcome: Number of High-risk Conditions Per Participant: Unmatched Participants
Description: High risk conditions included cancer, cerebrovascular or peripheral vascular disease, chronic lung disease, chronic liver disease, cystic fibrosis, dementia, diabetes, disability, heart conditions, HIV, hypertension, immunocompromised state(primary immunodeficiencies, prolonged use of corticosteroids or other immunosuppressive medications, and other immunocompromised state), mental health conditions(mood disorder or schizophrenia), overweight or obesity, physical inactivity, pregnancy(current or recent), sickle cell disease or thalassemia, smoking (current or former), solid organ or blood stem cell transplant, substance use disorder, tuberculosis. Index date=date of first COVID-19 diagnosis. Data was reported for unmatched participants, they were further sub-grouped on basis of outcome of COVID-19: eligible for absence from work, short term disability, long term disability. These sub-groups were not mutually exclusive; some participants might be represented in more than one category.
Time Frame: as for outcome 17
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: High-risk conditions per participant
Arm/Group | Unmatched Treated: Absence Eligibility | Unmatched Untreated: Absence Eligibility | Unmatched Treated: Short-term Disability | Unmatched Untreated: Short-term Disability | Unmatched Treated: Long-term Disability | Unmatched Untreated: Long-term Disability
Number analyzed (Participants) | 1931 | 9092 | 20076 | 90459 | 20336 | 94818
High-risk conditions per participant | 1.5 (1.2) | 1.5 (1.2) | 1.5 (1.2) | 1.4 (1.2) | 1.4 (1.2) | 1.4 (1.2)

24. Primary Outcome: Number of High-risk Conditions Per Participant: Matched Participants
Description: High risk conditions included cancer, cerebrovascular or peripheral vascular disease, chronic lung disease, chronic liver disease, cystic fibrosis, dementia, diabetes, disability, heart conditions, HIV, hypertension, immunocompromised state (primary immunodeficiencies, prolonged use of corticosteroids or other immunosuppressive medications, and other immunocompromised state), mental health conditions (mood disorder or schizophrenia), overweight or obesity, physical inactivity, pregnancy(current or recent), sickle cell disease or thalassemia, smoking (current or former), solid organ or blood stem cell transplant, substance use disorder, tuberculosis. Index date=date of first COVID-19 diagnosis. Data was reported for matched participants, they were further sub-grouped on basis of outcome of COVID-19: eligible for absence from work, short term disability, long term disability. These sub-groups were not mutually exclusive; some participants might be represented in more than one category.
Time Frame: as for outcome 17
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: High-risk conditions per participant
Arm/Group | Matched Untreated: Absence Eligibility | Matched Treated: Absence Eligibility | Matched Treated: Short-term Disability | Matched Untreated: Short-term Disability | Matched Treated: Long-term Disability | Matched Untreated: Long-term Disability
Number analyzed (Participants) | 1909 | 1909 | 20065 | 20065 | 20318 | 20318
High-risk conditions per participant | 1.5 (1.2) | 1.4 (1.2) | 1.5 (1.2) | 1.4 (1.2) | 1.4 (1.2) | 1.4 (1.2)

25. Primary Outcome: Number of Participants According to COVID-19 Vaccination Status: Unmatched Participant
Description: Number of participants with >=1 claim for a COVID-19 vaccination during the pre-period was reported in this outcome measure. Index date was the date of first COVID-19 diagnosis. In this outcome measure, data was reported for unmatched participants, they were further sub-grouped on the basis of outcome of COVID-19: eligible for absence from work, eligible for short term disability and eligible for long term disability. These sub-groups were not mutually exclusive; some participants might be represented in more than one category.
Time Frame: as for outcome 17
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Unmatched Treated: Absence Eligibility | Unmatched Untreated: Absence Eligibility | Unmatched Treated: Short-term Disability | Unmatched Untreated: Short-term Disability | Unmatched Treated: Long-term Disability | Unmatched Untreated: Long-term Disability
Number analyzed (Participants) | 1931 | 9092 | 20076 | 90459 | 20336 | 94818
Participants | 397 | 2101 | 4689 | 21611 | 4847 | 22478

26. Primary Outcome: Number of Participants According to COVID-19 Vaccination Status: Matched Participant
Description: Number of participants with >=1 claim for a COVID-19 vaccination during the pre-period was reported in this outcome measure. Index date was the date of first COVID-19 diagnosis. In this outcome measure, data was reported for matched participants, they were further sub-grouped on the basis of outcome of COVID-19: eligible for absence from work, eligible for short term disability and eligible for long term disability. These sub-groups were not mutually exclusive; some participants might be represented in more than one category.
Time Frame: as for outcome 17
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Matched Treated: Absence Eligibility | Matched Untreated: Absence Eligibility | Matched Treated: Short-term Disability | Matched Untreated: Short-term Disability | Matched Treated: Long-term Disability | Matched Untreated: Long-term Disability
Number analyzed (Participants) | 1909 | 1909 | 20065 | 20065 | 20318 | 20318
Participants | 391 | 297 | 4685 | 3761 | 4844 | 3845

27. Primary Outcome: Number of Participants With One or More Prior Hospitalization: Unmatched Participants
Description: Prior hospitalization indicated participants who had one or more inpatients visits in the pre-period. Index date was the date of first COVID-19 diagnosis. In this outcome measure, data was reported for unmatched participants, they were further sub-grouped on the basis of outcome of COVID-19: eligible for absence from work, eligible for short term disability and eligible for long term disability. These sub-groups were not mutually exclusive; some participants might be represented in more than one category.
Time Frame: as for outcome 17
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Unmatched Treated: Absence Eligibility | Unmatched Untreated: Absence Eligibility | Unmatched Treated: Short-term Disability | Unmatched Untreated: Short-term Disability | Unmatched Treated: Long-term Disability | Unmatched Untreated: Long-term Disability
Number analyzed (Participants) | 1931 | 9092 | 20076 | 90459 | 20336 | 94818
Participants | 41 | 291 | 421 | 2969 | 407 | 3096

28. Primary Outcome: Number of Participants With One or More Prior Hospitalization: Matched Participants
Description: Prior hospitalization indicated participants who had one or more inpatients visits in the pre-period. Index date was the date of first COVID-19 diagnosis. In this outcome measure, data was reported for matched participants, they were further sub-grouped on the basis of outcome of COVID-19: eligible for absence from work, eligible for short term disability and eligible for long term disability. These sub-groups were not mutually exclusive; some participants might be represented in more than one category.
Time Frame: as for outcome 17
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Matched Treated: Absence Eligibility | Matched Untreated: Absence Eligibility | Matched Treated: Short-term Disability | Matched Untreated: Short-term Disability | Matched Treated: Long-term Disability | Matched Untreated: Long-term Disability
Number analyzed (Participants) | 1909 | 1909 | 20065 | 20065 | 20318 | 20318
Participants | 37 | 31 | 419 | 444 | 406 | 432

29. Primary Outcome: Number of Participants With One or More Prior Emergency Room (ER) Visit: Unmatched Participants
Description: Prior ER visit indicates participants who had one or more ER visits in pre-period. Index date was the date of first COVID-19 diagnosis. In this outcome measure, data was reported for unmatched participants, they were further sub-grouped on the basis of outcome of COVID-19: eligible for absence from work, eligible for short term disability and eligible for long term disability. These sub-groups were not mutually exclusive; some participants might be represented in more than one category.
Time Frame: as for outcome 17
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Unmatched Treated: Absence Eligibility | Unmatched Untreated: Absence Eligibility | Unmatched Treated: Short-term Disability | Unmatched Untreated: Short-term Disability | Unmatched Treated: Long-term Disability | Unmatched Untreated: Long-term Disability
Number analyzed (Participants) | 1931 | 9092 | 20076 | 90459 | 20336 | 94818
Participants | 287 | 1884 | 2746 | 16507 | 2772 | 17760

30. Primary Outcome: Number of Participants With One or More Prior Emergency Room (ER) Visit: Matched Participants
Description: Prior ER visit indicates participants who had one or more ER visits in pre-period. Index date was the date of first COVID-19 diagnosis. In this outcome measure, data was reported for matched participants, they were further sub-grouped on the basis of outcome of COVID-19: eligible for absence from work, eligible for short term disability and eligible for long term disability. These sub-groups were not mutually exclusive; some participants might be represented in more than one category.
Time Frame: as for outcome 17
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study. This outcome measure was planned to be reported for matched participants (treated and untreated). Here, "Overall Number of Participants Analyzed (N)" signifies the numbers which were matched/ adjusted based on pre-defined characteristics among actual enrolled population and was a pseudo population, hence these numbers are different from unmatched population (actual enrolled population).
Measure: Count of Participants; unit: Participants
Arm/Group | Matched Treated: Absence Eligibility | Matched Untreated: Absence Eligibility | Matched Treated: Short-term Disability | Matched Untreated: Short-term Disability | Matched Treated: Long-term Disability | Matched Untreated: Long-term Disability
Number analyzed (Participants) | 1909 | 1909 | 20065 | 20065 | 20318 | 20318
Participants | 283 | 285 | 2738 | 2720 | 2770 | 2742

31. Primary Outcome: Number of Participants With Presence of Any Absence Records: Matched Participants
Description: Number of participants with presence of any absence records was reported in this outcome measure. Index date was the date of first COVID-19 diagnosis.
Time Frame: as for outcome 15
Population: Analysis population included all eligible participants whose data were included and observed in this study. This outcome measure was planned to be reported for matched participants (treated and untreated) who were eligible for absence from work due to COVID-19. Here, "N"=numbers which were matched/ adjusted based on pre-defined characteristics among actual enrolled population and was a pseudo population, hence these numbers are different from unmatched population (actual enrolled population).
Measure: Count of Participants; unit: Participants
Arm/Group | Matched Treated: Absence Eligibility | Matched Untreated: Absence Eligibility
Number analyzed (Participants) | 1909 | 1909
Participants | 1255 | 1331

32. Primary Outcome: Mean Number of Absence Days Per Participant Per Month (PPPM): Matched Participants
Description: In this outcome measure mean number of absence days PPPM was reported. Index date was the date of first COVID-19 diagnosis.
Time Frame: as for outcome 15
Population: Analysis population included all eligible participants whose data were included and observed in this study. Outcome measure was planned to be reported for matched participants(treated and untreated) who were eligible for absence. "N"=participants evaluable for outcome measure and numbers which were matched/ adjusted based on pre-defined characteristics among actual enrolled population and was a pseudo population, hence numbers are different from unmatched population (actual enrolled population).
Measure: Mean (Standard Deviation); unit: Days PPPM
Arm/Group | Matched Treated: Absence Eligibility | Matched Untreated: Absence Eligibility
Number analyzed (Participants) | 1255 | 1331
Days PPPM | 16.5 (19.0) | 17.8 (19.9)

33. Primary Outcome: Number of Participants According to Type for Absence Claim: Matched Participants
Description: Absence days was reported by absence type: sick, disability and recreational absence. Sick, disability and recreational absence were the leaves which participants took during the study period. Sick absence referred to the time away from work due to an employee's own illness or medical condition, this may be also used for bereavement, caring for a family member with a serious health condition, adoption-related medical needs. Disability absence was recorded when an employee was unable to work due to a short-term or long-term disability. Recreational absence referred to the time off taken for non-medical, personal reasons, such as vacation, personal leave, leisure, or wellness days. Index date was the date of first COVID-19 diagnosis. One participant may have more than one type of absence claim.
Time Frame: as for outcome 15
Population: as for outcome 32
Measure: Count of Participants; unit: Participants
Arm/Group | Matched Treated: Absence Eligibility | Matched Untreated: Absence Eligibility
Number analyzed (Participants) | 1255 | 1331
Participants
  Sick absence | 587 | 624
  Disability absence | 92 | 100
  Recreational absence | 1215 | 1286

34. Primary Outcome: Mean Cost of Absence Days: Matched Participants
Description: Estimated sum of wages associated with absence days was calculated as daily wage multiplied by absence days was reported PPPM in this outcome measure. Index date was the date of first COVID-19 diagnosis.
Time Frame: as for outcome 15
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: United states (US) Dollars PPPM
Arm/Group | Matched Treated: Absence Eligibility | Matched Untreated: Absence Eligibility
Number analyzed (Participants) | 1255 | 1331
United states (US) Dollars PPPM | 434 (504) | 468 (519)

35. Primary Outcome: Number of Participants With Any Short Term Disability (STD) Claim: Matched Participants
Description: Number of participants with presence of any STD claim was reported in this outcome measure. Index date was the date of first COVID-19 diagnosis.
Time Frame: as for outcome 15
Population: Analysis population included all eligible participants whose data were included and observed in this study. This outcome measure was planned to be reported for matched participants (treated and untreated) who were eligible STD. Here, "N"=numbers which were matched/ adjusted based on pre-defined characteristics among actual enrolled population and was a pseudo population, hence these numbers are different from unmatched population (actual enrolled population).
Measure: Count of Participants; unit: Participants
Arm/Group | Matched Treated: Short-term Disability | Matched Untreated: Short-term Disability
Number analyzed (Participants) | 20065 | 20065
Participants | 1343 | 1848

36. Primary Outcome: Mean Number of STD Days PPPM: Matched Participants
Description: In this outcome measure mean number of STD days PPPM was reported. Index date was the date of first COVID-19 diagnosis.
Time Frame: as for outcome 15
Population: Analysis population included all eligible participants whose data were included and observed in this study. Outcome measure was planned to be reported for matched participants(treated and untreated) who were eligible for STD."N"=participants evaluable for this outcome measure and numbers which were matched/ adjusted based on pre-defined characteristics among actual enrolled population and was a pseudo population, hence numbers are different from unmatched population (actual enrolled population).
Measure: Mean (Standard Deviation); unit: Days PPPM
Arm/Group | Matched Treated: Short-term Disability | Matched Untreated: Short-term Disability
Number analyzed (Participants) | 1343 | 1848
Days PPPM | 0.4 (2.2) | 0.5 (2.4)

37. Primary Outcome: Number of Participants According to Reason for STD Claim: Matched Participants
Description: Reasons for STD were classified as COVID-19 related or non-COVID-19 related or missing/unknown. Index date was the date of first COVID-19 diagnosis.
Time Frame: as for outcome 15
Population: Analysis population included all eligible participants whose data were included and observed in this study. Outcome measure was planned to be reported for matched participants(treated and untreated)who were eligible for STD. "N"=participants evaluable for this outcome measure and numbers which were matched/ adjusted based on pre-defined characteristics among actual enrolled population and was a pseudo population, hence numbers are different from unmatched population (actual enrolled population).
Measure: Count of Participants; unit: Participants
Arm/Group | Matched Treated: Short-term Disability | Matched Untreated: Short-term Disability
Number analyzed (Participants) | 1343 | 1848
Participants
  COVID-19-related | 220 | 327
  Not COVID-19-related | 1086 | 1462
  Missing/unknown | 37 | 59

38. Primary Outcome: Mean Cost of STD Days: Matched Participants
Description: Estimated sum of wages associated with absence days STD claim was calculated as 70 percentage (%) of daily wage multiplied by STD days was reported PPPM in this outcome measure. Index date was the date of first COVID-19 diagnosis.
Time Frame: as for outcome 15
Population: as for outcome 37
Measure: Mean (Standard Deviation); unit: United states (US) Dollars PPPM
Arm/Group | Matched Treated: Short-term Disability | Matched Untreated: Short-term Disability
Number analyzed (Participants) | 1343 | 1848
United states (US) Dollars PPPM | 84 (452) | 108 (506)

39. Primary Outcome: Number of Participants With Any Long Term Disability (LTD) Claim: Matched Participants
Description: Number of participants with presence of any LTD claim was reported in this outcome measure. Index date was the date of first COVID-19 diagnosis.
Time Frame: as for outcome 15
Population: Analysis population included all eligible participants whose data were included and observed in this study. This outcome measure was planned to be reported for matched participants (treated and untreated) who were eligible for LTD. Here, "N" signifies the numbers which were matched /adjusted based on pre-defined characteristics among actual enrolled population and was a pseudo population, hence these numbers are different from unmatched population (actual enrolled population).
Measure: Count of Participants; unit: Participants
Arm/Group | Matched Treated: Long-term Disability | Matched Untreated: Long-term Disability
Number analyzed (Participants) | 20318 | 20318
Participants | 50 | 74

40. Primary Outcome: Mean Number of LTD Days PPPM: Matched Participants
Description: In this outcome measure mean number of LTD days PPPM was reported. Index date was the date of first COVID-19 diagnosis.
Time Frame: as for outcome 15
Population: Analysis population included all eligible participants whose data were included and observed in this study. Outcome measure was planned to be reported for matched participants(treated and untreated)who were eligible for LTD. "N"=participants evaluable for this outcome measure and numbers which were matched/ adjusted based on pre-defined characteristics among actual enrolled population and was a pseudo population, hence numbers are different from unmatched population (actual enrolled population).
Measure: Mean (Standard Deviation); unit: Days PPPM
Arm/Group | Matched Treated: Long-term Disability | Matched Untreated: Long-term Disability
Number analyzed (Participants) | 50 | 74
Days PPPM | 0.02 (0.61) | 0.04 (0.78)

41. Primary Outcome: Number of Participants According to Reason for LTD Claim: Matched Participants
Description: Reasons for LTD were classified as COVID-19 related or non-COVID-19 related or missing/unknown. Index date was the date of first COVID-19 diagnosis.
Time Frame: as for outcome 15
Population: as for outcome 40
Measure: Count of Participants; unit: Participants
Arm/Group | Matched Treated: Long-term Disability | Matched Untreated: Long-term Disability
Number analyzed (Participants) | 50 | 74
Participants
  COVID-19-related | 1 | 1
  Not COVID-19-related | 33 | 58
  Missing/unknown | 16 | 15

42. Primary Outcome: Mean Cost of LTD Days: Matched Participants
Description: Estimated sum of wages associated with absence days LTD claim was calculated as 70 percent (%) of daily wage multiplied by LTD days was reported PPPM in this outcome measure. Index date was the date of first COVID-19 diagnosis.
Time Frame: as for outcome 15
Population: as for outcome 40
Measure: Mean (Standard Deviation); unit: United states (US) Dollars PPPM
Arm/Group | Matched Treated: Long-term Disability | Matched Untreated: Long-term Disability
Number analyzed (Participants) | 50 | 74
United states (US) Dollars PPPM | 4 (126) | 7 (164)

ADVERSE EVENTS:
Time Frame: Not applicable as adverse events and all-cause mortality were not planned to be evaluated/ monitored for the study
Description: Due to non-interventional nature of the study and nature of data sources, the minimum criteria for reporting an adverse event (i.e., identifiable participant, identifiable reporter, a suspect product, and event) could not be met, hence adverse events were not planned to be assessed or monitored (thus at risk appears "0").
Arm/Group | Unmatched Treated Cohort | Unmatched Untreated Cohort
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-29): https://cdn.clinicaltrials.gov/large-docs/93/NCT07072793/Prot_SAP_000.pdf